CLINICAL TRIAL: NCT06180161
Title: Effects of Multidomain Intervention on Cognitive Function in Community-dwelling Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202300820B0
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention grou[ (Experimental): Behavioral: multidomain intervention Dosage: a 2-hour session once a week for 12 weeks. Each multidomain intervention session includes 1 hour of combined physical (balance, strength and aerobic exercises) and cognitive (attention, memory, calculation, visual-spatial ability, processing speed and executive function) training and 1 hour of risk factor prevention and management strategies (nutrition, chronic disease management, oral health, fall prevention and transportation safety, psychosocial factors and sleep).
  Interventions: Behavioral: multidomain intervention
- control group (No Intervention): Waiting for 12 weeks (waiting-list control group)

INTERVENTIONS:
Behavioral: multidomain intervention — "Integrating exercise cognitive training with nutrition, chronic disease management, oral health, fall prevention, traffic safety, psychosocial well-being, and sleep to enhance the effectiveness of improving cognitive function in the elderly community."
  Arms: intervention grou[

SUMMARY:
The aging population has contributed to an increase in cognitive decline. To mitigate the rise in the dementia population, it is crucial to prevent cognitive decline in older adults with normal functioning, subjective cognitive decline (SCD), and mild cognitive impairment (MCI). Maintaining cognitive abilities as early as possible is essential for improved overall health and quality of life.

Healthcare for the elderly should focus on strengthening health promotion related to aging factors, such as cognitive function, mobility, nutrition, chronic disease management, oral health, fall prevention, transportation safety, psychosocial factors, and sleep. Additionally, as the etiology of dementia is multifactorial, numerous studies have been devoted to multidomain intervention, targeting multiple factors and domains in combination to enhance functions. The cumulative or synergistic effects of multidomain have garnered significant attention for their effectiveness in improving or maintaining the function of the elderly.

Therefore, this study aims to evaluate the effects of multidomain intervention, including combined physical and cognitive training, nutrition, chronic disease management, oral health, fall prevention, transportation safety, psychosocial factors, and sleep, on cognitive function in community-dwelling older adults.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years old
2. Mini-Mental State Examination (MMSE) score > 20 (Folstein et al., 1975), able to follow instructions and participate in activities
3. With self-reported or caregiver-reported memory or cognitive-related problems
4. No diagnosis of any type of dementia

Exclusion Criteria:

1. Unstable medical condition that would prevent safe participation in exercise training (e.g., myocardial infarction, heart failure, recent cardiac surgery, severe asthma, concomitant neurological disorders, or joint deformities)
2. Participation in other studies
3. Inability to provide informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change scores of Montreal Cognitive Assessment (MoCA) | baseline, after the intervention 12 weeks
  The MoCA is used to assess general cognitive functions. It examines several cognitive domains with a total score of 30 and higher values indicate better cognitive functions. The MoCA has been shown to be a valid and promising tool to evaluate the global cognitive function in patients with stroke. The psychometric properties of MoCA are good to excellent for patients with cerebrovascular diseases.
Change scores of Color Trials Test (CTT) | baseline, after the intervention 12 weeks
  The CTT is used to access executive function. For Part 1, the respondent uses a pencil to rapidly connect circles numbered 1-25 in sequence. For Part 2, the respondent rapidly connects numbered circles in sequence, but alternates between pink and yellow. The length of time to complete each trial is recorded, along with qualitative features of performance indicative of brain dysfunction, such as near-misses, prompts, number sequence errors, and color sequence errors.
Change scores of Stroop test | baseline, after the intervention 12 weeks
  The participants will be tested under congruent and incongruent conditions. In the congruent condition, the participant will name the color ink of a word which is consistent with the written color name; whereas in the incongruent condition the participant will name the color ink differs from the written color name. The time to complete the task will be calculated for each condition. Shorter time and less error indicate better inhibitory control.
Change scores of Digit symbol substitution test (DSST) of Wechsler Adult Intelligence Scale-Third Edition (WAIS-III) | baseline, after the intervention 12 weeks
  The DSST is used to assess information processing speed. The DSST involves a key consisting of the numbers 1-9, each paired with a unique, easy-to-draw symbol such as a "V", "+" or ">". Participant is asked to match symbols to numbers and copy the symbols into spaces within a 120-second timeframe. More correct symbols indicate better information processing speed.
Change scores of Spatial span test (SST) of Wechsler Memory Scale-Third Edition (WMS-III) | baseline, after the intervention 12 weeks
  The SST is used to assess working memory. Participants watch the assessor tap a sequence of blocks and are asked to tap it in order or reverse-order. More correct responses indicate better working memory.
Change scores of the Everyday Cognition scales-12 items (ECog-12) | baseline, after the intervention 12 weeks
  The ECog-12 is developed as an informant-rated report of cognitively mediated functional abilities in older adults. The ECog-12 asks participants to rate their current ability to perform cognitively mediated daily tasks related to everyday memory, language, visuospatial abilities, and executive functions compared with their ability to do the same task 10 years ago. Items are rated on a scale of 1-4, with 1 = Better or no change and 4 = Consistently much worse. The global, executive, and memory ECog-12 sub-domain scores are generated by averaging over the component items (sum of items/number of items) to maintain a range of 1 to 4 (with higher scores reflecting greater self-reported SCD).
Change scores of Timed up and go (TUG) | baseline, after the intervention 12 weeks
  The TUG assesses the dynamic balance ability and functional mobility. The participants will be required to stand up from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. The time to complete the TUG test has been shown to be a good indicator to detect potential fallers in frail elderly. The test-retest reliability of TUG on individuals with cognitive impairment is excellent.
Change scores of Short Physical Performance Battery (SPPB) | baseline, after the intervention 12 weeks
  The SPPB is an objective assessment tool for global physical function. The SPPB is a group of measures that combines the results of the side-by-side, semi-tandem and tandem stands (10 s), and 4 m walk test at a comfortable speed, and 5 quickly sit to stand. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability.
Change scores of the Lawton-Brody Instrumental Activities of Daily Living Scale (Lawton-Brody IADL Scale) | baseline, after the intervention 12 weeks
  The Lawton-Brody IADL Scale is a self-report questionnaire used to assess an individual's ability to perform instrumental activities of daily living, which are considered more complex and socially oriented than basic activities of daily living (BADLs). The scale is structured in a way that assigns points for each activity based on the individual's level of independence. The scoring may range from 0 to a maximum score, with a higher total score indicating a higher level of independence.
Change scores of 15-item Geriatric Depression Scale (GDS-15) | baseline, after the intervention 12 weeks
  The GDS-15 is a self-report scale used to evaluate depressive state in elderly individuals. The score range is 0-15, and a score of 5 or greater is taken as a possible indicator of depression.
Change scores of Community Integration Questionnaire (CIQ) | baseline, after the intervention 12 weeks
  The CIQ is designed to assess social participation, including home integration, social integration, and productive activity. The instrument consists of 15 items and can be completed by self-report or with the assistance of a family member or caregiver familiar with the person's health status and social activities.
Change scores of World Health Organization Quality of Life-brief version (WHOQOL-BREF) Taiwan Version | baseline, after the intervention 12 weeks
  The WHOQOL-BREF Taiwan version is used to access subjective quality of life. As with the standard WHOQOL-BREF questionnaires, the WHOQOL-BREF Taiwan version is simplified from the WHOQOL long form for Taiwan. For cross-cultural comparison, the first 26 items are the same as the standard WHOQOL-BREF, which is developed from global studies. In addition to the 26 items, applied the psychometric criteria proposed by the WHOQOL Group to select two more items from each of the two new facets to form the WHOQOL-BREF Taiwan version using data from the same 1,068 subjects. The selection process used for national items is described in the Results section. Thus, the WHOQOL-BREF Taiwan version contains 28 items classified into the same four domains as the standard WHOQOL-BREF. The scale administration and scoring procedures are the same as for the WHOQOL long form except that the facet score is based on only one item.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memotial Hospital, Taoyuan District, Taiwan